CLINICAL TRIAL: NCT04074018
Title: Clinical, Kinematic and Quality-of-life Related Impacts of Two Rehabilitation Programs in Chronic Peripheral Facial Paresis: a Randomized Control Trial.
Brief Title: Impacts of Two Rehabilitation Programs on Chronic Peripheral Facial Paresis
Acronym: VISAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K170105J
Record Dates: First submitted 2019-07-23; First posted 2019-08-29 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Facial Palsy; Self-rehabilitation; Quality of Life; Motor Recovery
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups, using computerized randomization, for the duration of the study in each center.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Self-rehabilitation guided program with investigator PMR specialist
  Interventions: Other: Self-rehabilitation program
- Control group (Active Comparator): Conventional rehabilitation with a speech therapist or physiotherapist specialized in facial rehabilitation
  Interventions: Other: Conventional rehabilitation program

INTERVENTIONS:
Other: Self-rehabilitation program — facial self-rehabilitation for a duration of 6 months
  Arms: Experimental group
Other: Conventional rehabilitation program — Conventional facial rehabilitation for a duration of 6 months
  Arms: Control group

SUMMARY:
Introduction: Peripheral facial paresis (PFP) is a very common disease of various etiologies affecting average adults with no predominance of sex. In 70% of cases, motor recovery is rapid and complete, but in 30% of early PFP, motor symptoms such as paresis and/or abnormal movements (synkinesis, contractures and/or spasms) can live on and jeopardize patients quality of life at medium and even long term. Concerning therapeutic interventions, the rehabilitation patient care of PFP is often restricted to the early stage. A recent randomized controlled study showed that early rehabilitation had a positive impact on motor recovery, specifically in severe motor grades, and could also accelerate time of recovery without exacerbating synkinesis. At chronic stage of the pathology, there is no controlled study testing the effect of motor rehabilitation when deficiencies are often considered as fitted and permanents.

Objective: It is well known in other domains that intensive motor strengthening increases cerebral plasticity in general, and particularly that of sensorimotor command. The main hypothesis of the study is that motor strengthening even at chronic stage of PFP could increase motor function and decrease abnormal motor movements through a self-rehabilitation motor program. The main objective is thus to compare the clinical, kinematic and quality-of-life related impacts of two different rehabilitation programs on motor recovery in unilateral PFP at chronic stage (i.e. at least 1 year after injury): a self-rehabilitation program guided by Physical Medicine and Rehabilitation (PMR) therapist versus facial rehabilitation involving physiotherapist or speech therapist specialized in facial rehabilitation. The main evaluation criterion is the evolution of the Sunnybrook Facial Grading Scale composite score between Day0 (before rehabilitation) and Day180 (after 6 months of facial rehabilitation).

Method: National, Randomized simple blind controlled study, in two parallel groups: Both program have to be realized daily for 6 months (Day1 to Day180). The population is made of adults with unilateral PFP at chronic stage i.e. at least 1 year from injury. Evaluations and follow-up of patients will be accomplished in a single center: Service de Rééducation Neurolocomotrice de l'Hôpital Mondor in Créteil (France).

ELIGIBILITY:
Inclusion Criteria:

* Age > 17 yo;
* Ambulatory patient;
* Motivation to participate to a rehabilitative facial program for six months;
* Patient consent to shaving (men) and no makeup (women) in order not to hamper evaluations the morning of the 4 visits of the study ;
* Signed informed consent;
* Affiliation to asocial security scheme.

Exclusion Criteria:

* Peripheral facial paresis of evolving tumoral etiology;
* Medical history of botulinum toxin injections in facial muscles during the last 6 months preceding inclusion or injections planned during the study;
* Medical history of facial surgery in the last two years preceding inclusion or planned during the study;
* Medical history of facial reanimation surgery needing specific rehabilitation (V-VII or XII-VII anastomosis or muscle transfer);
* Medical history of medical aesthetic facial treatments (hyaluronic acid/ lipofilling/laser/bracing wires) in the preceding two years before inclusion or planned during the study;
* Recurrent PFP;
* Implication in other research interventional protocol dealing with aesthetical aspect of the face or with PFP;
* Intercurrent pathology impeding the realization of the rehabilitation program during the study;
* Cognitive, mental or psychiatric troubles impeding the realization of the rehabilitation program or the capacity to attend both evaluations and follow-up consultations;
* Tutorship or guardianship patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change of Composite score of the Sunnybook Facial Grading System | Day 0 and Day 180
  estimation of resting symmetry (score 0 to 20), symmetry at voluntary movement (score 20 to 100) and synkinesis (score 0 to 15) composite score = symmetry at voluntary movement - resting symmetry - synkinesis from Day 0 to Day 180. (Ross et al. 1996, PMID: 8649870)

CONTACTS AND LOCATIONS:
Overall Officials: Marjolaine BAUDE, MD, Principal Investigator — APHP CHU HENRI MONDOR
Locations (3):
- France (3):
  - Centre Hospitalier Intercommunal de Créteil, Créteil, Val De Marne
  - Hôpital Henri Mondor, Créteil, Val De Marne
  - Hôpital Saint-Joseph, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baude M, Guihard M, Gault-Colas C, Benichou L, Coste A, Meningaud JP, Schmitz D, Natella PA, Audureau E, Gracies JM. Guided Self-rehabilitation Contract vs conventional therapy in chronic peripheral facial paresis: VISAGE, a multicenter randomized controlled trial. BMC Neurol. 2023 Apr 10;23(1):148. doi: 10.1186/s12883-023-03096-8. PMID 37038105